CLINICAL TRIAL: NCT06336083
Title: Family Screening for Internal Carotid Diaphragm Dysplasia (carotid WEB): a Doppler Ultrasound Study
Brief Title: Familial Form of Carotid Web: a Doppler Ultrasound Study
Acronym: Family-WEB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RC31/23/0618
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Carotid Web
Keywords: echography doppler; carotid web; inheritance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doppler ultrasound (Experimental): First degree relatives of patient with diagnosed carotid web will receive an echography doppler of the carotid arteries and answer questionnaires
  Interventions: Procedure: Doppler ultrasound

INTERVENTIONS:
Procedure: Doppler ultrasound — Participants will receive doppler ultrasound of the carotid arteries, and no other interventions studied

SUMMARY:
There is no evidence of familial forms of carotid web. The aim of this study is to determine the prevalence of carotid web among relatives of patient with carotid web using carotid doppler ultrasound.

DETAILED DESCRIPTION:
Carotid web are rare, focal dysplasia of the internal carotid artery and a high risk causes of stroke in young adult. Natural history of these dysplasia remains poorly understood. High prevalence of carotid web among Afro-Caribbean population and the similarity between carotid web and fibromuscular dysplasia, suggest existence of genetic factors. But there has been to our knowledge no familial form of carotid web reported. The aim of this study is to determine the prevalence of carotid web among relatives of patients with carotid web using carotid duplex doppler ultrasound.

Researchers aim to test whether carotid web could be detected in relatives of patients with known carotid web, using duplex doppler ultrasound.

This is a pilot, transversal, single-center study performed at Toulouse University Hospital, France. From 30 carotid web cases aged under 65 (patients with previously known Carotid web, symptomatic or not) followed in neurology department, investigators aim to include 60 first-degree relatives younger than 65 years old. Included relatives will underwent carotid duplex doppler ultrasound to detect carotid web. The primary outcome is the prevalence of carotid web among relatives. Secondary outcomes include : Number of families with at least one relative who has been diagnosed with carotid web, number of relatives who has been diagnosed with carotid web per family, clinical characteristics of patients and morphological characteristics of carotid web.

ELIGIBILITY:
Inclusion Criteria:

Carotid Web index patients:

* Patients with carotid web confirmed by CT angiogram (CTA) of cervical arteries or digital substraction angiogram (DSA).
* At least one first degree relative aged younger than 65 years old.

Relatives patients :

- First degree relatives of patient with diagnosed carotid web.

Exclusion Criteria:

* Persons placed under judicial protection or under another protection status
* Pregnant or breastfeeding woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prevalence of carotid web by doppler ultrasound in first-degree relatives of patients with carotid web. | Inclusion day
  Number of first-degree relatives with at least one carotid web on doppler ultrasound.

SECONDARY OUTCOMES:
Description of the clinical characteristics of relatives with carotid web and their index case. | Inclusion day
  Clinical characteristics of relatives with a carotid web and index cases: age, sex, vascular risk factors, medical history, family history, current treatments, bilateral nature of the carotid web.
Description of the morphological characteristics of relatives with carotid web and their index case. | Inclusion day
  Morphological characteristics on doppler ultrasound of the carotid web in relatives and in index cases: length, width, echogenicity, hemodynamic impact.

CONTACTS AND LOCATIONS:
Overall Officials: Claire VILLEPINTE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No